CLINICAL TRIAL: NCT03012750
Title: Angiosome Perfusion After Tibial Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Ulrich Rother, Dr. med. Ulrich Rother, Principal Investigator, University Hospital Erlangen
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: SPY-Angiosome
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- foot perfusion (Experimental): intravenous application of indocyanine green in patients receiving tibial Bypass surgery
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Perioperative application of 0.1 mg ICG per kg Body weight

SUMMARY:
Microcirculation should be assessed before and after tibial bypass surgery by intraoperative fluorescence angiography. According to this, the direct and the indirect angiosomes should be compared according to the individual microcirculatory improvement.

DETAILED DESCRIPTION:
Only patients at CLI stage Rutherford IV to VI with the necessity of tibial Bypass surgery will be included. Macrocirculation is measured by the ankle-brachial index (ABI). In order to assess the skin microcirculation intraoperative fluorescence angiography is used (SPY Elite™, NOVADAQ, Canada). The alteration of microcirculation is compared in direct and indirect revascularized angiosomes by calculation of the fluorescence parameters Ingress (IN) and Ingress rate (InR). Clinical Follow-up investigations will be performed and the wound healing rate is compared between the different revascularization methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients at CLI Rutherford stages IV to VI
* Patients with necessity of tibial Bypass surgery

Exclusion Criteria:

* Allergy against indocyanine green
* Iodine allergy
* Contrast allergy
* Penicillin allergy
* Allergic diathesis
* Liver insufficiency
* Pregnancy
* Hyperthyreosis
* Pulmonary arterial hypertension

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the direct and indirect revascularized angiosomes of the foot on the Level of microcirculation (Parameter Ingress) | 12 months
  Comparison of the fluorescence parameter Ingress in the direct and indirect revascularized angiosome before and after tibial bypass surgery
Comparison of the direct and indirect revascularized angiosomes of the foot on the Level of microcirculation (Parameter Ingressrate) | 12 months
  Comparison of the fluorescence parameter Ingressrate in the direct and indirect revascularized angiosome before and after tibial bypass surgery

SECONDARY OUTCOMES:
Correlation of the wound healing rates with indirect and direct revascularization | 12 months

REFERENCES:
- [Derived] Rother U, Lang W, Horch RE, Ludolph I, Meyer A, Gefeller O, Regus S. Pilot Assessment of the Angiosome Concept by Intra-operative Fluorescence Angiography After Tibial Bypass Surgery. Eur J Vasc Endovasc Surg. 2018 Feb;55(2):215-221. doi: 10.1016/j.ejvs.2017.11.024. Epub 2018 Jan 3. PMID 29305093